CLINICAL TRIAL: NCT03631732
Title: A Phase 3b, Multicenter, Open-Label Study to Evaluate Switching From a Regimen of Two Nucleos(t)Ide Reverse Transcriptase Inhibitors (NRTI) Plus a Third Agent to a Fixed Dose Combination (FDC) of Bictegravir/Emtricitabine/Tenofovir Alafenamide (B/F/TAF), in Virologically-Suppressed, HIV-1 Infected African American Participants
Brief Title: Study to Evaluate Switching From a Regimen of Two Nucleos(t)Ide Reverse Transcriptase Inhibitors (NRTI) Plus a Third Agent to a Fixed Dose Combination (FDC) of Bictegravir/Emtricitabine/Tenofovir Alafenamide (B/F/TAF), in Virologically-Suppressed, HIV-1 Infected African American Participants
Acronym: BRAAVE 2020
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-380-4580
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Results first posted 2020-08-27 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- B/F/TAF (Experimental): Participants will receive B/F/TAF (50/200/25 mg) FDC tablet orally once daily for 48 weeks, without regard to food. At Week 48, participants who wish to continue on B/F/TAF will be given the option to receive B/F/TAF FDC for up to an additional 24 weeks or until they have access to B/F/TAF, whichever occurs first.
  Interventions: Drug: B/F/TAF
- Stay on Baseline Regimen (SBR)/ Delayed B/F/TAF (Active Comparator): Participants will stay on baseline regimen consisting of 2 NRTIs and a third agent (each taken as prescribed) for 24 weeks with a delayed switch to B/F/TAF (50/200/25 mg) FDC tablet administered orally, once daily until Week 48 without regard to food. At Week 48, participants who wish to continue on B/F/TAF will be given the option to receive B/F/TAF FDC for up to an additional 24 weeks or until they have access to B/F/TAF, whichever occurs first.
  Interventions: Drug: B/F/TAF; Drug: NRTIs; Drug: Third Agent

INTERVENTIONS:
Drug: B/F/TAF — 50/200/25 mg FDC tablets administered orally once daily without regard to food
  Other Names: Biktarvy®
Drug: NRTIs — The following NRTIs will be administered as prescribed until Week 24 without regard to food:
  abacavir (ABC), emtricitabine (FTC), lamivudine (3TC), tenofovir alafenamide (TAF), tenofovir disoproxil fumarate (TDF), zidovudine (ZDV or AZT)
  Arms: Stay on Baseline Regimen (SBR)/ Delayed B/F/TAF
Drug: Third Agent — Any one of the following third agents will be administered as prescribed. Protease inhibitors and EVG will be administered with the appropriate pharmacologic booster cobicistat or ritonavir. :
  * Non-nucleoside reverse transcriptase inhibitors (NNRTIs)
    * delavirdine (DLV)
    * efavirenz (EFV)
    * nevirapine (NVP)
    * rilpivirine (RPV)
    * doravirine (DOR)
  * Integrase inhibitors
    * dolutegravir (DTG)
    * elvitegravir (EVG)
    * raltegravir (RAL)
  * Protease inhibitors (PIs)
    * atazanavir (ATV)
    * darunavir (DRV)
    * lopinavir (LPV)
    * nelfinavir NFV)
    * saquinavir (SQV)
    * tipranavir (TPV)
  * Chemokine co-recptor 5 (CCR5) antagonist --maraviroc (MVC)
  Arms: Stay on Baseline Regimen (SBR)/ Delayed B/F/TAF

SUMMARY:
The primary objective of this study is to evaluate the efficacy of switching from a regimen of 2 nucleos(t)Ide reverse transcriptase inhibitors (NRTIs) and a third agent to a fixed dose combination (FDC) of bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) versus continuing their baseline regimen in HIV-1 infected, virologically suppressed African American participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Self-describes as Black, African American, or mixed race, including Black
* Currently receiving an antiretrovirals (ARV) regimen other than FDC of B/F/TAF that consists of any two NRTIs + allowed 3rd agent for ≥ 6 months
* Allowed 3rd agents include any FDA-approved INSTI, with the exception of bictegravir, any FDA-approved NNRTI with the exception of etravirine, protease inhibitors or the CCR5 antagonist, maraviroc
* If the baseline 3rd agent is dolutegravir, dosing other than 50 mg once daily is excluded
* Baseline regimens containing investigational drugs or > 2 classes of ARVs are not permitted, with the exception of the pharmacologic enhancers cobicistat (taken with elvitegravir or a PI), or ritonavir (taken with a PI)
* Have no documented or suspected resistance to INSTIs and no history of virologic failure on an INSTI containing regimen (2 consecutive HIV-1 RNA ≥ 50 copies/mL after achieving <50 copies/mL while on an INSTI-containing regimen)
* History of 1-2 thymidine analogue mutations (TAMs), M184V/I, and any other RT substitutions are allowed, with the following exceptions: History of 3 or more TAMs (M41L, D67N, K70R, L210W, T215F/Y, and K219Q/E/N/R), T69-insertions, or K65R/E/N in RT will be excluded
* Documented plasma HIV-1 RNA < 50 copies/mL during treatment with the baseline regimen for a minimum period of 6 months and at least the last two HIV-1 RNA measurements prior to the Screening visit
* HIV-1 RNA levels < 50 copies/mL at Screening
* Estimated glomerular filtration rate (eGFR) ≥ 50 mL/min according to the Cockcroft-Gault formula for creatinine clearance

Key Exclusion Criteria:

* History of 3 or more TAMs (M41L, D67N, K70R, L210W, T215F/Y, and K219Q/E/N/R),T69-insertions, or K65R/E/N in RT
* No desire to switch from current ARVs
* An opportunistic illness indicative of stage 3 HIV diagnosed within the 30 days prior to screening
* Participants experiencing decompensated cirrhosis (e.g., ascites, encephalopathy, or variceal bleeding)
* Have been treated with immunosuppressant therapies or chemotherapeutic agents within 3 months of study screening, or expected to receive these agents or systemic steroids during the study (eg, corticosteroids, immunoglobulins, and other immune- or cytokine-based therapies)
* Malignancy within 5 years of screening other than cutaneous Kaposi's sarcoma, completely resected non -melanoma skin cancer (basal cell carcinoma or non-invasive cutaneous squamous carcinoma), or completely resected carcinoma in-situ of the cervix (CIN 3) or anus (AIN 3). A prior malignancy treated with curative therapy and for which there has been no evidence of disease for at least five years prior to screening is allowed
* Current alcohol or substance use judged by the Investigator to potentially interfere with participant study compliance
* Active, serious infections (other than HIV-1 infection) requiring antibiotic or antifungal therapy within 30 days prior to Day 1
* Participation in any other clinical trial, including observational studies, without prior approval from the sponsor is prohibited while participating in this trial
* Any other clinical condition or prior therapy that, in the opinion of the Investigator, would make the participant unsuitable for the study or unable to comply with the dosing requirements
* Known hypersensitivity to FDC of B/F/TAF tablets, their metabolites, or formulation excipient
* Females who are pregnant (as confirmed by positive serum pregnancy test)
* Females who are breastfeeding
* Acute hepatitis in the 30 days prior to randomization
* Active tuberculosis infection.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2020-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (82):
- United States (82):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Alabama Medical Group, PC, Mobile, Alabama
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Ruane Clinical Research Group Inc., Los Angeles, California
  - Mills Clinical Research, Los Angeles, California
  - Highland Hospital- Alameda Health System, Oakland, California
  - Kaiser Permanente, Oakland, California
  - One Community Health, Sacramento, California
  - Kaiser Permanente, Sacramento, California
  - Kaiser Permanente, Department of Infectious Diseases, San Leandro, California
  - Whitman-Walker Health, Washington D.C., District of Columbia
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Dupont Circle Physician's Group, Washington D.C., District of Columbia
  - Washington Health Institute, Washington D.C., District of Columbia
  - Capital Medical Associates, PC, Washington D.C., District of Columbia
  - The GW Medical Faculty Associates, Washington D.C., District of Columbia
  - Midland Florida Clinical Research Center, LLC, DeLand, Florida
  - Therafirst Medical Center, Fort Lauderdale, Florida
  - Gary J. Richmond, M.D., P.A., Fort Lauderdale, Florida
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - AHF- The Kinder Medical Group, Miami, Florida
  - University of Miami School of Medicine Division of Infectious Disease, Miami, Florida
  - AIDS Healthcare Foundation - South Beach, Miami Beach, Florida
  - Orlando Immunology Center, Orlando, Florida
  - St. Joseph's Hospital Comprehensive Research Institute, Tampa, Florida
  - AIDS Research & Treatment Center of the Treasure Coast, Vero Beach, Florida
  - Triple O Research Institute, P.A., West Palm Beach, Florida
  - Emory Hospital Midtown Infectious Disease Clinic, Atlanta, Georgia
  - Atlanta ID Group, PC, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Infectious Disease Specialist of Atlanta, Decatur, Georgia
  - Mercer University, Department of Internal Medicine, Macon, Georgia
  - Chatham County Health Department, Savannah, Georgia
  - Howard Brown Health Center, Chicago, Illinois
  - NorthStar Medical Center, Chicago, Illinois
  - Indiana CTSI Clinical Research Center, Indianapolis, Indiana
  - University Medical Center- New Orleans (UMCNO), New Orleans, Louisiana
  - SLVHCS Building J, 7th floor, Outpatient Infectious Disease Clinic, New Orleans, Louisiana
  - CrescentCare Health, New Orleans, Louisiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - Claudia T. Martorell, MD, LLC d/b/a The Research Institute, Springfield, Massachusetts
  - Be Well Medical Center, Berkley, Michigan
  - Wayne State University- Integrative Bioscience Center, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - St. John Newland Medical Associates, Southfield, Michigan
  - Hennepin County Medical Center, Positive Care Clinic, Minneapolis, Minnesota
  - G.V. 'Sonny' Montgomery VAMC, Jackson, Mississippi
  - Southampton Clinical Research, St Louis, Missouri
  - Clinical: Saint Louis University, New Hope Clinic, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Southampton Healthcare, Inc., St Louis, Missouri
  - Huntridge Family Clinic, Las Vegas, Nevada
  - Prime Healthcare Services- St. Michael's LLC d/b/a Saint Michael's Medical Center, Newark, New Jersey
  - North Shore University Hospital/Division of Infectious Diseases, Manhasset, New York
  - Jacobi Medical Center, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - NC TraCS Institute-CTRC; University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - UT Physicians, Charlotte, North Carolina
  - Duke University Health System, Durham, North Carolina
  - East Carolina University, The Brody School of Medicine, ECU Adult Specialty Care, Greenville, North Carolina
  - Rosedale Infectious Diseases, Huntersville, North Carolina
  - AHF, Pensacola, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Perelman Center for Advanced Medicine at the Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Philadelphia FIGHT Community Health Centers, Philadelphia, Pennsylvania
  - Palmetto Health Richland, Columbia, South Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Central Texas Clinical Research, Austin, Texas
  - St. Hope Foundation, Bellaire, Texas
  - AIDS Arms, Inc. DBA Prism Health North Texas, Dallas, Texas
  - North Texas Infectious Diseases Consultants, P.A., Dallas, Texas
  - Tarrant County Infectious Disease Associates, Fort Worth, Texas
  - Therapeutic Concepts, PA, Houston, Texas
  - Thomas Street Health Center, Houston, Texas
  - Research Access Network, Houston, Texas
  - The Crofoot Research Center, INC (dba Gordon E. Crofoot MD PA), Houston, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Community Health Care, Hilltop Medical Clinic, Tacoma, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Result] Andreatta K, D'Antoni ML, Chang S, Parvangada A, Martin R, Blair C, et al. Preexisting Resistance and Week 48 Virologic Outcomes after Switching to B/F/TAF in African American Adults With HIV [Presentation]. IDWeek Virtual; 2020b 21-25 October.
- [Result] Hagins D, Kumar P, Saag M, Wurapa AK, Brar I, Berger D, Osiyemi O, Hileman CO, Ramgopol M, McDonald C, Blair C, Andreatta K, Collins SE, Brainard D, Martin H. Week-48 Outcomes From the BRAAVE 2020 Study: a Randomized Switch to B/F/TAF in African-American Adults With HIV, IDWeek 2020, October 21-25. Abstract 1046.
- [Result] Andreatta K, D'Antoni ML, Chang S, Martin R, Blair C, Collins SE, et al. Preexisting Resistance and B/F/TAF Switch Efficacy in African Americans [Poster 509]. Conference on Retroviruses and Opportunistic Infections (CROI); 2020b 08-11 March; Boston, MA.
- [Result] Hagins D, Kumar P, Saag M, Wurapa AK, Brar I, Berger D, Osiyemi O, Hileman CO, Ramgopol M, McDonald C, Blair C, Andreatta K, Collins SE, Brainard D, Martin H. Randomized Switch to B/F/TAF in African American Adults with HIV. Conference on Retroviruses and Opportunistic Infections 2020, March 7-11, Boston MA. Abstract 2979.
- [Result] Hagins D, Kumar P, Saag M, Wurapa AK, Brar I, Berger D, Osiyemi O, Hileman CO, Ramgopal MN, McDonald C, Blair C, Andreatta K, Collins SE, Brainard DM, Martin H; BRAAVE2020 Investigators. Switching to Bictegravir/Emtricitabine/Tenofovir Alafenamide in Black Americans With HIV-1: A Randomized Phase 3b, Multicenter, Open-Label Study. J Acquir Immune Defic Syndr. 2021 Sep 1;88(1):86-95. doi: 10.1097/QAI.0000000000002731. PMID 34397746

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study centers in the United States. The first participant was screened on 28 August 2018. The last study visit occurred on 19 August 2020.
Pre-assignment Details: The following NRTIs & 3rd agents were allowed:
  NRTIs:abacavir, emtricitabine, lamivudine, tenofovir alafenamide, tenofovir disoproxil fumarate, zidovudine;
  3rd agents:delavirdine,efavirenz, nevirapine, rilpivirine,dolutegravir, elvitegravir,raltegravir, doravirine, atazanavir, darunavir, lopinavir, nelfinavir, saquinavir, tipranavir, maraviroc
Groups:
- B/F/TAF: Participants received bictegravir /emtricitabine/tenofovir alafenamide (B/F/TAF) (50/200/25 mg) fixed dose combination (FDC) tablet orally once daily for 48 weeks, without regard to food. At Week 48, participants who wished to continue on B/F/TAF were given the option to receive B/F/TAF FDC for up to an additional 24 weeks or until they had access to B/F/TAF, whichever occurred first.
- Stay on Baseline Regimen (SBR)/ Delayed B/F/TAF: Participants stayed on baseline regimen consisting of 2 nucleos(t)Ide reverse transcriptase inhibitors (NRTIs) and a third agent (each taken as prescribed) for 24 weeks with a delayed switch to B/F/TAF (50/200/25 mg) FDC tablet administered orally, once daily until Week 48 without regard to food. At Week 48, participants who wished to continue on B/F/TAF were given the option to receive B/F/TAF FDC for up to an additional 24 weeks or until they had access to B/F/TAF, whichever occurred first.
Period: Randomized Phase Up to Week 24
Arm/Group | B/F/TAF | Stay on Baseline Regimen (SBR)/ Delayed B/F/TAF
Started | 331 | 165
Completed | 324 | 163
Not Completed | 7 | 2
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrew Consent | 1 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Randomized but not treated | 1 | 0
Period: B/F/TAF Treatment Phase (After Week 24)
Arm/Group | B/F/TAF | Stay on Baseline Regimen (SBR)/ Delayed B/F/TAF
Started | 319 (5 participants completed 24 weeks of the study, but did not receive study treatment after Week 24.) | 163
Completed | 303 | 158
Not Completed | 16 | 5
Not completed — Lost to Follow-up | 6 | 1
Not completed — Withdrew Consent | 3 | 3
Not completed — Adverse Event | 4 | 1
Not completed — Death | 1 | 0
Not completed — Investigator's discretion | 1 | 0
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who were randomized into the study and had received at least 1 dose of study treatment (either B/F/TAF or baseline regimen on Day 1).
Groups:
- B/F/TAF: Participants received B/F/TAF (50/200/25 mg) FDC tablet orally once daily for 48 weeks, without regard to food. At Week 48, participants who wished to continue on B/F/TAF were given the option to receive B/F/TAF FDC for up to an additional 24 weeks or until they had access to B/F/TAF, whichever occurred first.
- Stay on Baseline Regimen/ Delayed B/F/TAF: Participants stayed on baseline regimen consisting of 2 NRTIs and a third agent (each taken as prescribed) for 24 weeks with a delayed switch to B/F/TAF (50/200/25 mg) FDC tablet administered orally, once daily until Week 48 without regard to food. At Week 48, participants who wished to continue on B/F/TAF were given the option to receive B/F/TAF FDC for up to an additional 24 weeks or until they had access to B/F/TAF, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | B/F/TAF | Stay on Baseline Regimen/ Delayed B/F/TAF | Total
Number analyzed (Participants) | 330 | 165 | 495
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (12.3) | 48 (12.2) | 47 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 55 | 156
  Male | 229 | 110 | 339
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 5 | 20
  Not Hispanic or Latino | 315 | 160 | 475
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Black or African American | 285 | 154 | 439
  Native Hawaiian or Pacific Islander | 0 | 0 | 0
  White | 0 | 0 | 0
  Other | 45 | 11 | 56
HIV-1 RNA Category [Count of Participants; unit: Participants]
  < 50 copies/mL | 325 | 163 | 488
  ≥ 50 copies/mL | 5 | 2 | 7
CD4+ Cell Count [Mean (Standard Deviation); unit: cells/µL] | 765 (313.4) | 757 (323.0) | 763 (316.3)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Had HIV-1 RNA ≥ 50 Copies/mL at Week 24 as Defined by the US FDA-Defined Snapshot Algorithm: Full Analysis Set
Description: The percentage of participants who had HIV-1 RNA ≥ 50 copies/mL at Week 24 was analyzed using the snapshot algorithm, which defined a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 24
Population: Participants in the Full Analysis Set [included all participants who were randomized into the study, and had received at least 1 dose of study treatment (either B/F/TAF or baseline regimen on Day 1), and did not have pre-existing integrase strand transfer inhibitor resistance-associated mutations (based on historical data)] in B/F/TAF and SBR groups were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- B/F/TAF: Participants received B/F/TAF (50/200/25 mg) FDC tablet orally once daily for 48 weeks, without regard to food.
- Stay on Baseline Regimen (SBR): Participants stayed on baseline regimen consisting of 2 NRTIs and a third agent (each taken as prescribed) for 24 weeks administered orally once daily.
Arm/Group | B/F/TAF | Stay on Baseline Regimen (SBR)
Number analyzed (Participants) | 328 | 165
percentage of participants | 0.6 [0.1 to 2.2] | 1.8 [0.4 to 5.2]
Statistical Analysis 1: Comparison: B/F/TAF vs Stay on Baseline Regimen (SBR); Test type: Non-Inferiority — B/F/TAF is non-inferior to SBR if the upper bound of the 2-sided 95% confidence interval (CI) of the difference between treatment groups [B/F/TAF - SBR] in the percentage of participants with HIV-1 RNA ≥ 50 copies/mL is less than 6% (i.e., a margin of 6% is applied to non-inferiority assessment); Difference in percentages = -1.2, 95% CI 2-sided [-4.8 to 0.9] — Differences in percentages of participants with HIV-1 RNA >= 50 copies/mL between treatment groups and 95% CI were calculated based on exact method
Statistical Analysis 2: Comparison: B/F/TAF vs Stay on Baseline Regimen (SBR); Test type: Superiority; p = 0.3399, Fisher Exact

2. Secondary Outcome: Percentage of Participants Who Had HIV-1 RNA ≥ 50 Copies/mL at Week 48 as Defined by the US FDA-Defined Snapshot Algorithm: Full Analysis Set
Description: The percentage of participants who had HIV-1 RNA ≥ 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defined a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status. By Week 48, participants in B/F/TAF had received 48 weeks of treatment with B/F/TAF, while those in the Delayed B/F/TAF group had received only 24 weeks of treatment with B/F/TAF.
Time Frame: Week 48
Population: Participants in the Full Analysis Set in the B/F/TAF and the Delayed B/F/TAF groups with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Delayed B/F/TAF: Participants in SBR group who switched to B/F/TAF group at Week 24 received B/F/TAF (50/200/25 mg) FDC tablet orally, once daily from Week 24 until Week 48 without regard to food. At Week 48, participants who wished to continue on B/F/TAF were given the option to receive B/F/TAF FDC for up to an additional 24 weeks or until they had access to B/F/TAF, whichever occurred first.
Arm/Group | B/F/TAF | Delayed B/F/TAF
Number analyzed (Participants) | 328 | 163
percentage of participants | 0.9 [0.2 to 2.6] | 0 [0.0 to 2.2]

3. Secondary Outcome: Percentage of Participants Who Had HIV-1 RNA < 50 Copies/mL at Week 24 as Defined by the US FDA-Defined Snapshot Algorithm: Full Analysis Set
Description: The percentage of participants who had HIV-1 RNA < 50 copies/mL at Week 24 was analyzed using the snapshot algorithm, which defined a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 24
Population: Participants in the Full Analysis Set in the B/F/TAF and SBR groups were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | B/F/TAF | Stay on Baseline Regimen (SBR)
Number analyzed (Participants) | 328 | 165
percentage of participants | 96.3 [93.7 to 98.1] | 94.5 [89.9 to 97.5]
Statistical Analysis 1: Comparison: B/F/TAF vs Stay on Baseline Regimen (SBR); Test type: Non-Inferiority — B/F/TAF is non-inferior to SBR if the lower bound of the 2-sided 95% CI of the difference between treatment groups [B/F/TAF - SBR] in the percentage of participants with HIV-1 RNA < 50 copies/mL is greater than -10% (i.e., a margin of 10% is applied to non-inferiority assessment); Difference in percentages = 1.8, 95% CI 2-sided [-2.0 to 6.8] — Differences in percentages of participants with HIV-1 RNA < 50 copies/mL between treatment groups and 95% CI were calculated based on exact method
Statistical Analysis 2: Comparison: B/F/TAF vs Stay on Baseline Regimen (SBR); Test type: Superiority; p = 0.3532, Fisher Exact

4. Secondary Outcome: Percentage of Participants Who Had HIV-1 RNA < 50 Copies/mL at Week 24 as Defined by the US FDA-Defined Snapshot Algorithm: Week 24 Per Protocol Analysis Set
Description: as for outcome 3
Time Frame: Week 24
Population: Participants in the Week 24 Per Protocol Analysis Set [included all participants who were randomized into the study and had received at least 1 dose of study treatment (either B/F/TAF or baseline regimen on Day 1), and had not committed any major protocol violation, including the violation of key entry criteria] in the B/F/TAF and SBR groups were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | B/F/TAF | Stay on Baseline Regimen (SBR)
Number analyzed (Participants) | 306 | 148
percentage of participants | 99.3 [97.7 to 99.9] | 98.0 [94.2 to 99.6]
Statistical Analysis 1: Comparison: B/F/TAF vs Stay on Baseline Regimen (SBR); Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Difference in percentages = 1.4, 95% CI 2-sided [-1.0 to 5.3] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: B/F/TAF vs Stay on Baseline Regimen (SBR); Test type: Superiority; p = 0.3356, Fisher Exact

5. Secondary Outcome: Percentage of Participants Who Had HIV-1 RNA < 50 Copies/mL at Week 48 as Defined by the US FDA-Defined Snapshot Algorithm: Full Analysis Set
Description: The percentage of participants who had HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defined a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status. By Week 48, participants in B/F/TAF had received 48 weeks of treatment with B/F/TAF, while those in the Delayed B/F/TAF group had received only 24 weeks of treatment with B/F/TAF.
Time Frame: Week 48
Population: Participants in the Full Analysis Set in the B/F/TAF and the Delayed B/F/TAF groups with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | B/F/TAF | Delayed B/F/TAF
Number analyzed (Participants) | 328 | 163
percentage of participants | 94.5 [91.5 to 96.7] | 96.9 [93.0 to 99.0]

6. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 24: Full Analysis Set
Description: The analysis includes values up to 1 day after permanent discontinuation of study treatment.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set in the B/F/TAF and SBR groups with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | B/F/TAF | Stay on Baseline Regimen (SBR)
Number analyzed (Participants) | 319 | 156
cells/uL | 13 (209.3) | 1 (171.2)
Statistical Analysis 1: Comparison: B/F/TAF vs Stay on Baseline Regimen (SBR); Test type: Other; p = 0.5618, ANOVA; P-value was calculated from ANOVA model with treatment as a fixed effect; Difference in LSM = 11, 95% CI 2-sided [-27 to 49] — Difference in LSM (Least square mean) and its 95% C.I. was calculated from ANOVA model with treatment as a fixed effect

7. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 24: Week 24 Per Protocol Analysis Set
Description: The analysis includes values up to 1 day after permanent discontinuation of study treatment.
Time Frame: Baseline to Week 24
Population: Participants in the Week 24 Per Protocol Analysis Set in the B/F/TAF and SBR groups with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | B/F/TAF | Stay on Baseline Regimen (SBR)
Number analyzed (Participants) | 305 | 144
cells/uL | 13 (210.1) | 4 (171.3)
Statistical Analysis 1: Comparison: B/F/TAF vs Stay on Baseline Regimen (SBR); Test type: Other; p = 0.6632, ANOVA; P-value was calculated from ANOVA model with treatment as a fixed effect; Difference in LSM = 9, 95% CI 2-sided [-31 to 48] — Difference in LSM and its 95% C.I. was calculated from ANOVA model with treatment as a fixed effect

8. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 48: Full Analysis Set
Description: The analysis includes values up to 1 day after permanent discontinuation of study treatment. By Week 48, participants in B/F/TAF had received 48 weeks of treatment with B/F/TAF, while those in the Delayed B/F/TAF group had received only 24 weeks of treatment with B/F/TAF.
Time Frame: Baseline to Week 48
Population: Participants in the Full Analysis Set in the B/F/TAF and the Delayed B/F/TAF groups with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | B/F/TAF | Delayed B/F/TAF
Number analyzed (Participants) | 309 | 159
cells/uL | 7 (188.6) | -8 (159.2)

9. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant administered a medicinal product, which did not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and/or unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A treatment-emergent adverse event was defined as any adverse event with onset date on or after the study treatment start date and no later than 30 days after the study drug stop date; or any adverse event leading to study drug discontinuation.
Time Frame: First B/F/TAF dose date up to Week 72 plus 30 days
Population: The B/F/TAF (BVY) Safety Analysis Set included all participants who were randomized into the study and received at least 1 dose of BVY study drug.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF | Delayed B/F/TAF
Number analyzed (Participants) | 330 | 163
percentage of participants | 83.3 | 69.3

10. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Graded Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as values that increase at least one toxicity grade from baseline. The most severe graded abnormality from all tests was counted for each participant. Severity grades were defined by 'Gilead Grading Scale for Severity of AEs and Laboratory Abnormalities'.
Time Frame: First B/F/TAF dose date up to Week 72 plus 30 days
Population: Participants in the BVY Safety Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF | Delayed B/F/TAF
Number analyzed (Participants) | 329 | 163
percentage of participants | 87.8 | 80.4

ADVERSE EVENTS:
Time Frame: Adverse Events: First B/F/TAF dose date up to Week 72 plus 30 days. All-Cause Mortality: Randomization up to Week 72 plus 30 days.
Description: The Safety Analysis Set included all participants who were randomized into the study and had received at least 1 dose of study treatment (either B/F/TAF or baseline regimen on Day 1).
  All-Cause Mortality: The All Randomized Analysis Set included all participants who were randomized into the study.
Groups:
- B/F/TAF up to Week 24: Participants received B/F/TAF (50/200/25 mg) FDC tablet orally once daily for 24 weeks, without regard to food.
- SBR up to Week 24: Participants stayed on baseline regimen consisting of 2 NRTIs and a third agent (each taken as prescribed) for 24 weeks administered orally once daily.
- B/F/TAF After Week 24: Participants received B/F/TAF (50/200/25 mg) FDC tablet orally once daily from Week 24 to Week 48, without regard to food. At Week 48, participants who wished to continue on B/F/TAF were given the option to receive B/F/TAF FDC for up to an additional 24 weeks or until they had access to B/F/TAF, whichever occurred first.
Arm/Group | B/F/TAF up to Week 24 | SBR up to Week 24 | B/F/TAF After Week 24 | Delayed B/F/TAF
All-Cause Mortality (participants affected / at risk) | 1/331 | 0/165 | 2/319 | 0/163
Serious Adverse Events (participants affected / at risk) | 13/330 | 7/165 | 20/319 | 7/163
Other Adverse Events (participants affected / at risk) | 38/330 | 13/165 | 53/319 | 26/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B/F/TAF up to Week 24 (N=330) | SBR up to Week 24 (N=165) | B/F/TAF After Week 24 (N=319) | Delayed B/F/TAF (N=163)
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 2 | 0
Complication associated with device (General disorders) | 0 | 0 | 0 | 1
Anal abscess (Infections and infestations) | 1 | 1 | 0 | 0
Anorectal infection (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Burn infection (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Covid-19 (Infections and infestations) | 0 | 0 | 3 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0 | 0
Neurosyphilis (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0
Lacunar infarction (Nervous system disorders) | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Vertebral artery dissection (Nervous system disorders) | 0 | 0 | 1 | 0
Bipolar I disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0
Homicidal ideation (Psychiatric disorders) | 1 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 2 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | B/F/TAF up to Week 24 (N=330) | SBR up to Week 24 (N=165) | B/F/TAF After Week 24 (N=319) | Delayed B/F/TAF (N=163)
Diarrhoea (Gastrointestinal disorders) | 11 | 5 | 4 | 9
Syphilis (Infections and infestations) | 4 | 1 | 18 | 7
Upper respiratory tract infection (Infections and infestations) | 20 | 6 | 17 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 2 | 16 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (4):
  • Study Protocol (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/32/NCT03631732/Prot_000.pdf
  • Statistical Analysis Plan: Week 24 Analysis (2019-08-30): https://cdn.clinicaltrials.gov/large-docs/32/NCT03631732/SAP_001.pdf
  • Statistical Analysis Plan: Final Analysis (2020-11-16): https://cdn.clinicaltrials.gov/large-docs/32/NCT03631732/SAP_002.pdf
  • Statistical Analysis Plan: Week 48 Analysis (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/32/NCT03631732/SAP_003.pdf